CLINICAL TRIAL: NCT05945797
Title: Can Deep Common Bile Duct Cannulation Time During Endoscopic Retrograde Cholangiopancreatography Be Shortened by Dexamethasone
Brief Title: Effects of Dexamethasone on Common Bile Duct Cannulation Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gujranwala medical college District Headquarters Hospital, Gujranwala (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2023-06-11; First posted 2023-07-14 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Common Bile Duct Diseases; Common Bile Duct Calculi; Common Bile Duct Stricture; Common Bile Duct Neoplasms; Common Bile Duct Dilatation
Keywords: ERCP, Steroids, Dexamethasone, CBD cannulation time
MeSH Terms: conditions — Common Bile Duct Diseases; Gallstones; Common Bile Duct Neoplasms | interventions — Dexamethasone; Steroids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexa Arm (Experimental): Experimental arm patients will be receiving 2 ml (4mg) of dexamenthasone prior to undergoing ERCP.
  Interventions: Drug: Dexamethasone 4mg
- NS Arm (Placebo Comparator): Placebo arm patients will be receiving 2 ml of normal saline prior to undergoing ERCP.
  Interventions: Drug: Dexamethasone 4mg

INTERVENTIONS:
Drug: Dexamethasone 4mg — An injection of 4mg of dexamethasone will be given to patients approximately 2 to 4 hours prior to the procedure of ERCP.
  Other Names: steroids

SUMMARY:
The main aim of this clinical trial is to evaluate the effects of dexamethasone on common bile duct cannulation time during endoscopic retrograde cholangiopancreatography (ERCP) in patients with biliary pathologies. The study will also study the effects of dexamethasone on total procedure time and total fluoroscopy time during ERCP.

Participants will be divided into two groups, treatment group and placebo group. Patients in treatment group will receive dexamethasone and those in placebo group will be given normal saline before undergoing ERCP. The results in both groups will be compared to determine the effects of dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years or above
* Both genders, male and female patients

Exclusion Criteria:

* Age younger than 18 years or below
* Pregnant females
* Pre existing stent in CBD or pancreatic duct
* Previous history of ERCP
* Patients with billroth II surgery
* Anatomical abnormalities
* Lack of competence in patients
* Roux en Y gastric bypass
* Patients with contra indications for steroids like DM

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
Shortening of CBD cannulation time | CBD cannulation time will be calculated from the start of the procedure (0 minutes) till complete CBD cannulation has been achieved through catheter and confirmed by fluoroscopy or procedure abandoned if unsuccessful cannulation by 30 minutes.
  To determine the effects of dexamethasone on shortening of CBD cannulation time

CONTACTS AND LOCATIONS:
Overall Officials: Najam us Sehar Saeed, FCPS-Gastro, Study Chair — GMC-DHQ Hospital, Gujwanala, Pakistan
Locations (1):
- Gujranwala Medical College Hospital, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sherman S, Lehman GA. Endoscopic retrograde cholangiopancreatography, endoscopic sphincterotomy and stone removal, and endoscopic biliary and pancreatic drainage. In: Yamada T, et al. (eds.) Text book of gastroenterology. 3rd edn. Philadelphia: Lippincott, Williams & Wilkins ; 1999: 2718 - 2746
- [Background] Wehrmann T, Schmitt T, Stergiou N, Caspary WF, Seifert H. Topical application of nitrates onto the papilla of Vater: manometric and clinical results. Endoscopy. 2001 Apr;33(4):323-8. doi: 10.1055/s-2001-13687. PMID 11315893
- [Background] Allescher HD, Neuhaus H, Hagenmuller F, Classen M. Effect of N-butylscopolamine on sphincter of Oddi motility in patients during routine ERCP--a manometric study. Endoscopy. 1990 Jul;22(4):160-3. doi: 10.1055/s-2007-1012829. PMID 2209497
- [Background] Sola-Bonada N, de Andres-Lazaro AM, Roca-Massa M, Bordas-Alsina JM, Codina-Jane C, Ribas-Sala J. [1.6% peppermint oil solution as intestinal spasmolytic in retrograde endoscopic cholangiopancreatography]. Farm Hosp. 2012 Jul-Aug;36(4):256-60. doi: 10.1016/j.farma.2011.08.003. Epub 2011 Dec 1. Spanish. PMID 22137159
- [Background] Devereaux BM, Lehman GA, Fein S, Phillips S, Fogel EL, Sherman S. Facilitation of pancreatic duct cannulation using a new synthetic porcine secretin. Am J Gastroenterol. 2002 Sep;97(9):2279-81. doi: 10.1111/j.1572-0241.2002.05982.x. PMID 12358245